CLINICAL TRIAL: NCT02444546
Title: Phase 1 Study of Replication Competent Reovirus (Reolysin®) in Combination With GM-CSF in Pediatric Patients With Relapsed or Refractory Brain Tumors
Brief Title: Wild-Type Reovirus in Combination With Sargramostim in Treating Younger Patients With High-Grade Relapsed or Refractory Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1472; NCI-2015-00665 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1472 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2015-05-01; First posted 2015-05-14 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Childhood Astrocytoma; Childhood Atypical Teratoid/Rhabdoid Tumor; Diffuse Intrinsic Pontine Glioma; Glioma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Brain Neoplasm; Recurrent Childhood Glioblastoma; Recurrent Childhood Medulloblastoma; Recurrent Primitive Neuroectodermal Tumor; Refractory Brain Neoplasm
MeSH Terms: conditions — Rhabdoid Tumor; Diffuse Intrinsic Pontine Glioma; Glioma; Oligodendroglioma; Astrocytoma; Medulloblastoma; Neuroectodermal Tumors, Primitive; Brain Neoplasms | interventions — sargramostim; Colony-Stimulating Factors; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sargramostim, wild-type reovirus) (Experimental): Patients receive sargramostim SC daily on days 1 and 2 and wild-type reovirus IV over 60 minutes on days 3-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sargramostim; Biological: Wild-type Reovirus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: Wild-type Reovirus — Given IV
  Other Names: Reolysin

SUMMARY:
This phase I trial studies the side effects and the best dose of wild-type reovirus (viral therapy) when given with sargramostim in treating younger patients with high grade brain tumors that have come back or that have not responded to standard therapy. A virus, called wild-type reovirus, which has been changed in a certain way, may be able to kill tumor cells without damaging normal cells. Sargramostim may increase the production of blood cells and may promote the tumor cell killing effects of wild-type reovirus. Giving wild-type reovirus together with sargramostim may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) and describe the toxicities of wild-type reovirus (Reolysin) when given once a day for three days following two days of treatment with sargramostim (GM-CSF).

SECONDARY OBJECTIVES:

I. To assess the safety, tolerability and adverse events in the patient population.

II. To assess the median overall survival time in this patient population. III. To assess the median progression free survival time in this patient population.

TERTIARY OBJECTIVES:

I. To determine whether there is a correlation between antibody responsiveness to the virus and a positive tumor response to Reolysin in patients who receive the virus following treatment with GM-CSF.

II. To determine whether there is a correlation between an increased number of circulating monocytes and a positive tumor response to Reolysin in patients who receive the virus following treatment with GM-CSF.

III. To explore the possible predictive value of monocyte numbers in response to Reolysin + GM-CSF therapy.

OUTLINE: This is a dose-escalation study of wild-type reovirus.

Patients receive sargramostim subcutaneously (SC) daily on days 1 and 2 and wild-type reovirus intravenously (IV) over 60 minutes on days 3-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of a high grade (grade 3 or 4) primary brain tumor either classified as a glioma (including astrocytoma, anaplastic oligodendroglioma and glioblastoma multiforme), medulloblastoma, atypical teratoid/rhabdoid tumor (AT/RT) or primitive neuroectodermal tumor (PNET)

  * Note: Patients with diffuse intrinsic pontine glioma (DIPG) are exempt from this confirmation of tumor if characteristic radiologic findings are noted on magnetic resonance imaging (MRI)
* Patients must have no known curative therapy available
* Evidence of tumor progression by MRI scan following radiation therapy or following the most recent anti-tumor therapy; note: patients who have had surgical treatment at recurrence are eligible if they had a resection with measurable residual disease on postoperative imaging or if there is imaging evidence of disease progression as compared to the first postoperative scan
* Measurable disease: measurable by gadolinium MRI scan
* Absolute neutrophil count (ANC) >= 750 /uL obtained =< 7 days prior to registration
* Absolute lymphocyte count (ALC) >= 250/uL obtained =< 7 days prior to registration
* Platelet count (PLT) >= 75,000 /uL without transfusions obtained =< 7 days prior to registration
* Hemoglobin >= 7.0 gm/dL obtained =< 7 days prior to registration
* Total bilirubin =< 1.5 times upper limit of institutional normal (ULN) for age obtained =< 7 days prior to registration
* Aspartate transaminase (AST) =< 3 times ULN for age obtained =< 7 days prior to registration
* Serum albumin >= 2 g/dL
* Creatinine =< 1.5 times ULN for age OR a creatinine clearance or glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2; obtained =< 7 days prior to registration
* Karnofsky or Lansky performance status (PS): performance status of >= 50 assessed within two weeks prior to registration; neurological deficits in patients must have been relatively stable for a minimum of 1 week prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Ability to understand and the willingness to provide written informed assent or consent
* Willing to return to enrolling institution for follow-up
* Immunosuppressants: patients must be receiving a stable or decreasing dose of dexamethasone for at least 1 week prior to start of therapy AND dexamethasone dose must be =< 0.1 mg/kg/day AND =< a total daily dose of 4 mg/day
* If patient has a clinically indicated surgery or biopsy at any time during treatment with Reolysin, a tissue sample will be collected for correlative research purposes
* Patient willing to provide mandatory blood samples for correlative research purposes; the inability to provide a blood sample or the lack of an available blood sample does not make the patient ineligible
* Negative urine or serum pregnancy test done =< 7 days prior to registration for females who are post-menarchal
* Patient agrees to use an acceptable form of contraception during the study and for up to 28 days after the last dose of Reolysin if patient or female partner is post-menarche; acceptable methods include 1) a double barrier method, such as condom and spermicide; 2) hormonal contraception methods, including pills, patches, rings, or injections except progestin-only containing pills (i.e., 'mini-pill'); 3) intrauterine device (non-progesterone T); 4) surgical methods such as a bilateral tubal ligation or a vasectomy; 5) abstinence
* Must be able to avoid direct contact with pregnant women, infants < 3 months of age and immunocompromised individuals while on study and for >= 3 weeks following the last dose of study agent administration; direct contact is defined as household contact, i.e., anyone living with the patient
* Life expectancy >= 3 months

Exclusion Criteria:

* Fetal and newborn toxicity: any of the following

  * Pregnant women
  * Nursing women
  * Males or post-menarchal females who are unwilling to employ adequate contraception throughout the duration of the study and for at least 4 weeks after treatment has ended
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection, including localized infections
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Any psychiatric illness/social situations that would limit compliance with study requirements
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known prior history of tuberculosis or positive purified protein derivative (PPD) test result
* Known prior history of human immunodeficiency virus (HIV)
* Administration of live vaccines =< 14 days prior to registration; note: patients may not receive any viral immunizations during the study and for 28 days after the last dose of Reolysin
* Prior history of any viral-based therapy
* Other concurrent chemotherapy, immunotherapy, radiotherapy, any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) or receiving any other investigational agent which would be considered as a treatment for the primary neoplasm:

  * Chemotherapy =< 3 weeks of registration
  * Nitrosoureas or mitomycin C =< 6 weeks of registration
  * Small molecule cell cycle inhibitors =< 2 weeks prior to registration
  * Immunotherapy =< 6 weeks prior to registration
  * Monoclonal antibodies =< 3 half-lives prior to registration
  * Radiation therapy

    * Last fraction of craniospinal irradiation or total body irradiation =< 3 months prior to registration or last fraction of focal irradiation to symptomatic metastatic sites =< 4 weeks prior to registration
  * Growth factors

    * Colony forming growth factors < 2 weeks prior to registration (i.e., filgrastim, sargramostim, erythropoietin)
    * Neulasta < 2 weeks prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06-21 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
MTD, based on the incidence of dose-limiting toxicity (DLT) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 | Up to 84 days
  MTD is the highest safely tolerated dose level where 1 of 6 patients experience DLT with the next higher dose having at least 2 patients out of a maximum of 6 patients experience DLT.

SECONDARY OUTCOMES:
Adverse event profile | Up to 5 years
  The number and severity of adverse events (overall, by dose level, by treatment received) will be tabulated and summarized. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Objective responses | Up to 5 years
  Objective responses will be summarized by descriptive summary statistics delineating complete and partial responses and stable and progressive disease.
Overall survival | Up to 5 years
  Will be summarized descriptively. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and relevant confidence intervals.
Time to progression | Will be summarized descriptively.
  Up to 5 years
Time to treatment failure | Up to 5 years
  Will be summarized descriptively. Time to treatment failure is defined as the time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient.
Time until any treatment-related toxicity | Up to 5 years
  Will be summarized descriptively.
Time until treatment-related grade 3+ toxicity | Up to 5 years
  Will be summarized descriptively.
Toxicity profile, assessed by CTCAE v4.0 | Up to 5 years
  Toxicity is defined as adverse events that are classified as possibly, probably, or definitely related to study treatment. Overall toxicity incidence and toxicity profiles by dose level, patient, and treatment will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of the analysis.

OTHER OUTCOMES:
Immunologic parameters | Up to 5 years
  For each of the immunologic parameters, a time series plot will be constructed. A grid reflecting the percent change from pre-treatment levels will be constructed. This grid will be analyzed to determine if the changes seen in each immunologic parameter differ between patients who response and those which do not respond.
Reovirus immune status | Up to 5 years
  The reovirus immune status will be correlated with objective response to analyze if the status is predictive of sargramostim plus wild-type reovirus therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bram, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States